CLINICAL TRIAL: NCT01620762
Title: A Double-Blind, Randomised, Placebo-Controlled Multi-Centre Field Study to Assess the Efficacy and Safety of Cat-PAD Peptide Immunotherapy in Cat Allergic Subjects
Brief Title: Phase III Cat-PAD Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: inVentiv Health Clinical (Other); Pharm-Olam International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP007
Record Dates: First submitted 2012-05-30; First posted 2012-06-15 (Estimated); Results first posted 2018-05-14 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Rhinoconjunctivitis
Keywords: Cat allergy; Rhinoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cat-Pad Treatment 1 (Experimental): Cat-PAD Treatment 1
  Interventions: Drug: Cat-PAD
- Cat-PAD Treatment 2 (Experimental): Cat-PAD Treatment regimen 2
  Interventions: Drug: Cat-PAD; Drug: Placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cat-PAD — 1 dose every 4 weeks
  Arms: Cat-PAD Treatment 2; Cat-Pad Treatment 1
Drug: Placebo — 1 dose every 4 weeks
  Arms: Cat-PAD Treatment 2; Placebo

SUMMARY:
The purpose of this study is to compare the treatment effect of two treatment regimens of Cat-PAD vs placebo and to evaluates the treatment effect of Cat-PAD on symptoms, rescue medication usage and Quality of Life.

ELIGIBILITY:
Inclusion Criteria

* Male or female, aged 12-65 years.
* Moderate to severe rhinoconjunctivitis on exposure to cats for at least 2 years.
* Subjects may optionally also have GINA Step 1 controlled asthma.
* Positive skin prick test to cat hair.
* Cat dander specific IgE ≥0.35 kU/L.

Exclusion Criteria

* Asthma falling under the GINA definitions "partly controlled" and "uncontrolled" or Steps 2 to 5.
* FEV1 <80% of predicted.
* Clinically significant confounding symptoms of allergy to seasonal allergens during the final evaluation period.
* Skin prick test 5 mm greater than the negative control to perennial allergens or animal dander (other than cat) which cannot be avoided during the study.
* Significant symptoms of another clinically relevant illness that is likely to affect scoring of rhinoconjunctivitis symptoms.
* Clinically relevant abnormalities detected on physical examination.
* History of severe drug allergy, severe angioedema or anaphylactic reaction to food.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1408 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold Nelson, MD, Principal Investigator — Jewish National Health
Locations (118):
- United States (52):
  - Rolling Hills Estates, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Wheat Ridge, Colorado
  - Eagle, Idaho
  - Meridian, Idaho
  - Chicago, Illinois
  - Evanston, Illinois
  - Forrest, Illinois
  - Normal, Illinois
  - Iowa City, Iowa
  - Overland Park, Kansas
  - Bangor, Maine
  - Brockton, Massachusetts
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Bozeman, Montana
  - Missoula, Montana
  - Bellevue, Nebraska
  - Fremont, Nebraska
  - Omaha, Nebraska
  - Ocean Township, New Jersey
  - Albuquerque, New Mexico
  - Corning, New York
  - Newburgh, New York
  - Fargo, North Dakota
  - Minot, North Dakota
  - Canton, Ohio
  - Cincinnati, Ohio
  - Middleburg Heights, Ohio
  - Sylvania, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Lake Oswego, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - Blue Bell, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Draper, Utah
  - Glen Allen, Virginia
  - South Burlington, Virginia
  - Warrenton, Virginia
  - Spokane, Washington
  - Greenfield, Wisconsin
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Canada (14):
  - Burlington, Ontario
  - Corruna, Ontario
  - Hamilton, Ontario
  - Kanata, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Niagara Falls, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Pointe-Claire, Quebec
  - Québec, Quebec
  - Trois-Rivières, Quebec
- Czechia (7):
  - Brnho
  - Čáslav
  - České Budějovice
  - Jablonec nad Nisou
  - Kutná Hora
  - Prague
  - Rychnov nad Kněžnou
- Germany (14):
  - Berlin
  - Bonn
  - Bramsche
  - Cologne
  - Hamburg
  - Heidelberg
  - Mönchengladbach
  - München
  - Münster
  - Neuss
  - Osnabrück
  - Wesel
  - Wiesbaden
  - Wuppertal
- Hungary (4):
  - Budapest
  - Csorna
  - Pécs
  - Tatabánya
- Poland (13):
  - Bydgoszcz
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Rzeszów
  - Tarnów
  - Warsaw
  - Wroclaw
  - Zabrze
  - Zawadzkie
- Russia (8):
  - Barnaul
  - Moscow
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Stavropol
  - Tomsk
  - Yekaterinburg
- Slovakia (3):
  - Bardejov
  - Martin
  - Poprad

RESULTS

PARTICIPANT FLOW:
Groups:
- Cat-PAD Treatment 1 (1 Course): Cat-PAD Treatment 1
  Cat-PAD: 1 dose every 4 weeks Placebo: 1 dose every 4 weeks
- Cat-PAD Treatment 2 (2 Courses): Cat-PAD Treatment regimen 2
  Cat-PAD: 1 dose every 4 weeks
Period: Overall Study
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment 2 (2 Courses) | Placebo
Started | 468 | 470 | 470
Completed | 420 | 412 | 417
Not Completed | 48 | 58 | 53
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Adverse Event | 9 | 5 | 2
Not completed — Withdrawal by Subject | 23 | 26 | 27
Not completed — Lost to Follow-up | 11 | 17 | 10
Not completed — Protocol deviation | 1 | 1 | 6
Not completed — Subject deterioration | 0 | 1 | 1
Not completed — Non-specified | 3 | 6 | 5
Not completed — Use of prohibted therapies | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment 2 (2 Courses) | Placebo | Total
Number analyzed (Participants) | 468 | 470 | 470 | 1408
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 29 | 32 | 90
  Between 18 and 65 years | 439 | 441 | 438 | 1318
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 301 | 317 | 317 | 935
  Male | 167 | 153 | 153 | 473
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 1 | 2 | 11
  Not Hispanic or Latino | 458 | 468 | 463 | 1389
  Unknown or Not Reported | 2 | 1 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Combined Score in Cat-PAD Treatment Groups Compared With Placebo
Description: The primary endpoint was the mean Combined Score (CS) measured over a 3 week period (52-54 weeks after randomisation) in the Cat-PAD treatment groups compared with the mean CS in the placebo group. A higher score indicated worse symptoms or greater use of medication and thus a low score indicated a better outcome.
  CS = Total Rhinoconjunctivitis Symptom Score (TRSS) + Rescue Medication Score (RMS). Eight symptoms are defined in the TRSS, 4 nasal symptoms: runny nose, sneezing; blocked nose, and itchy nose and 4 ocular symptoms: itchy eyes; watery eyes; red eyes and sore eyes. Each symptom was rated in severity on a score of 0-3 (0=absent, 3=severe) and the total was divided by the number of symptoms to provide an average score per symptom of 0-3.
  RMS was scored from 0 (no allergy rescue medication use per day) to 3 (at least one dose of systemic corticosteroid per day). The RMS score was not additive, and therefore the maximum RMS was 3 and the maximum CS was 6.
Time Frame: 52-54 weeks after randomisation
Population: Only those subjects in the intent to treat (ITT) population with data at the end of the study were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment 2 (2 Courses) | Placebo
Number analyzed (Participants) | 417 | 414 | 414
units on a scale | 1.04 (0.068) | 1.00 (0.068) | 1.05 (0.068)

2. Secondary Outcome: Mean TRSS
Description: Mean Total Rhinoconjunctivitis Symptom Score (TRSS) in Cat-PAD treatment groups compared with placebo.
  Eight symptoms are defined in the TRSS, 4 nasal symptoms: runny nose, sneezing; blocked nose, and itchy nose and 4 ocular symptoms: itchy eyes; watery eyes; red eyes, and sore eyes. Each symptom was rated in severity on a score of 0-3 (0. absent; 1. mild, barely noticeable; 2. moderate, annoying/troublesome; 3. severe, very annoying/very troublesome), therefore TRSS could range from 0 to 24. Higher TRSS reflected more severe symptom scores. Symptoms were scored daily for a period of approximately 3 weeks. 52-54 weeks after randomisation.
Time Frame: 52-54 weeks after randomisation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment 2 (2 Courses) | Placebo
Number analyzed (Participants) | 417 | 414 | 414
units on a scale | 5.67 (0.358) | 5.54 (0.356) | 5.87 (0.357)

3. Secondary Outcome: Mean Daily TNSS in Cat-PAD Compared With Placebo
Description: TNSS (Total nasal symptom score) was the sum of all the nasal symptom scores (runny nose; sneezing; blocked nose; itchy nose) and could range from 0 to 12. Higher TNSS reflected more severe symptoms.
  Subjects rated the severity of each symptom over the last 24 hours as follows: 0. absent; 1. mild, barely noticeable; 2. moderate, annoying/troublesome; 3. severe, very annoying/very troublesome. Symptoms were scored daily for a period of approximately 3 weeks. 52-54 weeks after randomisation.
Time Frame: 52-54 weeks after randomisation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment 2 (2 Courses) | Placebo
Number analyzed (Participants) | 417 | 414 | 414
units on a scale | 3.48 (0.197) | 3.36 (0.196) | 3.44 (0.196)

4. Secondary Outcome: Mean Daily TOSS in Cat-PAD Compared to Placebo
Description: Mean daily Total Ocular Symptom Score (TOSS) in Cat-PAD treatment groups compared to placebo groups
  TOSS was the sum of all the ocular symptom scores (itchy eyes; watery eyes; red eyes; sore eyes) and could range from 0 to 12. Higher TOSS reflected more severe symptoms.
  Subjects rated the severity of each symptom over the last 24 hours as follows: 0. absent; 1. mild, barely noticeable; 2. moderate, annoying/troublesome; 3. severe, very annoying/very troublesome. Symptoms were scored daily for a period of approximately 3 weeks. 52-54 weeks after randomisation.
Time Frame: 52-54 weeks after randomisation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment 2 (2 Courses) | Placebo
Number analyzed (Participants) | 417 | 414 | 414
units on a scale | 2.20 (0.179) | 2.19 (0.178) | 2.42 (0.179)

5. Secondary Outcome: Mean RMS in Cat-PAD Compared With Placebo
Description: Mean RMS (Rescue medication score) in Cat-PAD treatment groups compared with placebo groups.
  The use of rhinoconjunctivitis rescue medications was recorded by the subject on a daily basis just before bedtime for approximately 21 days, 52-54 weeks after randomisation and was scored based on a previously published system as follows: 0 = no allergy rescue medication used per day; 0.5 = at least one dose of antihistamine eye drops used per day; 1 = at least one dose of oral antihistamine used per day; 2 = at least one dose of intranasal corticosteroid used per day; 3 = at least one dose of systemic corticosteroid used per day. The score was according to the highest level of rescue medication used and was not additive.
Time Frame: 52-54 weeks after randomisation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment 2 (2 Courses) | Placebo
Number analyzed (Participants) | 417 | 414 | 414
units on a scale | 0.34 (0.038) | 0.31 (0.037) | 0.32 (0.037)

6. Secondary Outcome: Mean RQLQ Score in Cat-PAD Compared With Placebo
Description: The RQLQ (Rhinoconjunctivitis Quality of Life Questionnaire) was completed by subjects at the end of the study (52-54 weeks after randomisation).
  The RQLQ is a validated method of assessing quality of life and has 28 questions in seven domains (activity limitation, sleep problems, nasal symptoms, eye symptoms, non-nasal/eye symptoms, practical problems and emotional function). Subjects recalled how their rhinoconjunctivitis had been during the last week and responded to each question on a seven-point scale (0 = no impairment, 6 = maximum impairment). The questions were equally weighted, and the RQLQ score was the mean of the 28 questions and could range from zero to six.
Time Frame: 52-54 weeks after randomisation
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment 2 (2 Courses) | Placebo
Number analyzed (Participants) | 396 | 403 | 393
units on a scale | 1.26 (0.080) | 1.26 (0.079) | 1.25 (0.079)

7. Secondary Outcome: Number of Days With no Moderate or Severe TRSS Symptoms Without Rescue Medication Use
Description: The number of well days, i.e., days with no moderately or severely annoying symptoms and with no rescue medication used was calculated for all subjects over a period of approximately 21 days, 52-54 weeks after randomisation.
Time Frame: 52-54 week after randomisaiton
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment 2 (2 Courses) | Placebo
Number analyzed (Participants) | 417 | 414 | 414
days | 9.44 (0.56) | 10.11 (0.556) | 9.76 (0.557)

ADVERSE EVENTS:
Time Frame: Up to 52 weeks after randomisation
Description: The number of participants at risk for AEs and SAEs is for the safety population, one participant withdrew after randomisation but before receiving any treatment and is therefore included in the ITT population and therefore in the participant flow module but is not included in the safety population. The data presented reflects the data in the TLFs and as written in the Clinical Study Report.
Arm/Group | Cat-PAD Treatment 1 (1 Course) | Cat-PAD Treatment 2 (2 Courses) | Placebo
Serious Adverse Events (participants affected / at risk) | 11/467 | 13/470 | 9/470
Other Adverse Events (participants affected / at risk) | 298/467 | 299/470 | 305/470
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cat-PAD Treatment 1 (1 Course) (N=467) | Cat-PAD Treatment 2 (2 Courses) (N=470) | Placebo (N=470)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hydonephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cat-PAD Treatment 1 (1 Course) (N=467) | Cat-PAD Treatment 2 (2 Courses) (N=470) | Placebo (N=470)
Allergy to animal (Immune system disorders) | 9 (9) | 9 (11) | 11 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (26) | 18 (27) | 24 (26)
Orophayngeal pai (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 16 (20) | 16 (18)
Athma (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 14 (15) | 16 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (19) | 7 (13) | 11 (12)
Headache (Nervous system disorders) | 25 (78) | 39 (86) | 35 (76)
Injection site pruritus (General disorders) | 19 (51) | 13 (45) | 11 (41)
Injection site urticaria (General disorders) | 17 (95) | 9 (43) | 7 (41)
Pyrexia (General disorders) | 6 (6) | 12 (13) | 6 (7)
Nausea (Gastrointestinal disorders) | 9 (10) | 12 (12) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 6 (7) | 12 (15)
Toothache (Gastrointestinal disorders) | 1 (1) | 11 (12) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (20) | 9 (12) | 15 (20)
Athralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 12 (16) | 16 (16)
Nasopharyngitis (Infections and infestations) | 85 (124) | 87 (128) | 90 (127)
Upper respiratory tract infection (Infections and infestations) | 37 (48) | 34 (41) | 42 (60)
Sinusitis (Infections and infestations) | 21 (26) | 24 (29) | 23 (24)
Bronchitis (Infections and infestations) | 23 (27) | 23 (25) | 19 (21)
Pharyngitis (Infections and infestations) | 11 (11) | 18 (20) | 14 (17)
Influenza (Infections and infestations) | 9 (9) | 5 (5) | 19 (20)
Urinary tract infection (Infections and infestations) | 9 (11) | 12 (16) | 11 (13)
Tonsillitis (Infections and infestations) | 9 (11) | 10 (12) | 7 (7)
Rhinitis (Infections and infestations) | 8 (8) | 4 (5) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
To avoid disclosures that may affect the proprietary rights of the Sponsor, the Investigator agrees to allow Circassia the opportunity to review all manuscripts and abstracts 60 days prior to submission for publication. Circassia reserves the right to include the report of this study in any regulatory documentation or submission or in any informational materials.